CLINICAL TRIAL: NCT06807645
Title: Evaluating the Impact of Prefabricated Acrylic Splints on Premaxillary Stability in Alveolar Cleft Bone Graft Repairs: a Randomized Controlled Trial
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Majidah ALhussain, Principal Investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS3-3-8; CairoU (Other: University of Cairo)
Record Dates: First submitted 2025-01-24; First posted 2025-02-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Bilateral Complete Cleft Lip And/or Alveolus and Acrylic Splint, and; Maxillary Deficiency; Stability
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Intervention Model Description: Interventions
  All surgical procedures will be conducted under general anesthesia with nasotracheal intubation, and a first-generation cephalosporin will be administered as antibiotic prophylaxis prior to incision Bowder et al. (2021). Autogenous bone grafts will be harvested from the anterior iliac crest using a pediatric minimally invasive technique, involving a 2 cm skin incision made 1 cm lateral to the iliac crest, meticulously dissected to preserve soft tissue. pain management strategies will be employed postoperatively to ensure comprehensive pain control and enhance patient comfort throughout the recovery period.
  For the alveolar cleft repair, a sulcular incision will be made to develop full thickness mucoperiosteal advancement flaps extending into the cleft, with careful elevation of buccal
Masking Description: I have 2 group, partipant will have the intervention another no.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical Trial Intervention Description General Study Setup Objective: To compare the efficacy of us (Experimental): Clinical Trial Intervention Description General Study Setup Objective: To compare the efficacy of using a custom-made prefabricated acrylic splint versus no splint in maintaining premaxillary stability post-alveolar cleft repair.
  Primary Outcome: Premaxillary stability. Secondary Outcomes: Wound healing and complications. Intervention Details
  1. Common Procedures for Both Arms:
  Surgical Procedure: All surgical procedures will be conducted under general anesthesia with nasotracheal intubation.
  Antibiotic Prophylaxis: A first-generation cephalosporin will be administered prior to incision as per Bowder et al. (2021).
  Bone Graft Harvesting: Autogenous bone grafts will be harvested from the anterior iliac crest using a pediatric minimally invasive technique with a 2 cm skin incision 1 cm lateral to the iliac crest.
  Alveolar Cleft Repair:
  Incision and Flap Design: A sulcular incision will be made to develop full thickness mucoperiosteal advancement flaps extending into the cleft with care
  Interventions: Device: Clinical Trial Intervention Description General Study Setup Objective: To compare the efficacy of using a custom-made prefabricated acrylic splint versus no splint in maintaining premaxillary stabilit

INTERVENTIONS:
Device: Clinical Trial Intervention Description General Study Setup Objective: To compare the efficacy of using a custom-made prefabricated acrylic splint versus no splint in maintaining premaxillary stabilit — Clinical Trial Intervention Description General Study Setup Objective: To compare the efficacy of using a custom-made prefabricated acrylic splint versus no splint in maintaining premaxillary stability post-alveolar cleft repair.
  Primary Outcome: Premaxillary stability. Secondary Outcomes: Wound healing and complications. Intervention Details
  1. Common Procedures for Both Arms:
  Surgical Procedure: All surgical procedures will be conducted under general anesthesia with nasotracheal intubation.
  Antibiotic Prophylaxis: A first-generation cephalosporin will be administered prior to incision as per .
  Bone Graft Harvesting: Autogenous bone grafts will be harvested from the anterior iliac crest using a pediatric minimally invasive technique with a 2 cm skin incision 1 cm lateral to the iliac crest.
  Alveolar Cleft Repair:
  Incision and Flap Design: A sulcular incision will be made to develop full thickness mucoperiosteal advancement flaps extending into the cleft with caref

SUMMARY:
Rationale for conducting the research:

Bilateral alveolar clefts pose significant management challenges, with current treatments like autogenous bone grafting showing instability in up to 40% of cases within a year, risking graft failure and aesthetic issues . Prefabricated acrylic splints may offer a minimally invasive alternative, potentially improving bone graft outcomes and premaxillary stability, crucial for speech, feeding, and respiration. This study evaluates the efficacy of acrylic splinting versus traditional open healing, aiming to enhance patient outcomes and reduce healthcare costs associated with this congenital condition . This research underscores the need for evidence-based, minimally invasive treatments that can improve quality of life and guide clinical practices for managing bilateral alveolar clefts.

Review of literature:

The existing body of literature on bilateral alveolar clefts and their management reflects several inadequacies and gaps in the evidence base. Bilateral alveolar clefts present unique challenges that have not been fully addressed in the literature on cleft lip and palate management. Limited evidence suggests more focused research in this area. The prevailing treatment options for bilateral alveolar clefts predominantly involve surgical bone grafting procedures. These grafting techniques have shown varying success rates, with factors such as graft quality, surgical technique, and premaxillary stability influencing outcomes. However, the specific challenges posed by bilateral alveolar clefts have not been addressed comprehensively in the existing literature. While grafting procedures have undoubtedly improved the lives of countless patients, there remains a need for more targeted interventions that can enhance premaxillary stability and graft success, particularly in the context of bilateral alveolar clefts. The proposed use of prefabricated acrylic splints represents a novel and innovative approach to address these inadequacies. These splints are designed to provide consistent and reliable support to the premaxilla during the critical early phases of healing following grafting procedures. By minimizing premaxillary mobility, they have the potential to enhance graft success rates, improve premaxillary stability, and enhance the overall outcomes of bilateral alveolar cleft repairs.

Explanation for choice of comparators:

standard bone grafting without acrylic splints is considered the 'gold standard' for treating alveolar clefts. Using normal repair as the comparator allows for a clear assessment of the possible advantages and challenges of incorporating acrylic splints into existing best practices.

7. Objectives:

Aim of the Study The primary aim of this study is to assess the impact of prefabricated acrylic splints on premaxillary stability, soft tissue healing, and graft stability in patients with bilateral alveolar clefts.

Hypothesis:

Null Hypothesis (H0): Bilateral alveolar cleft patients who receive prefabricated acrylic splints have similar premaxillary stability, soft tissue healing, and graft stability.

Alternative Hypothesis (H1): Prefabricated acrylic splints improve premaxillary stability, soft tissue healing, and graft stability in bilateral alveolar cleft patients.

The above hypotheses are neutral and not biased. The study tests these hypotheses to obtain objective and evidence-based conclusions about prefabricated acrylic splints for bilateral alveolar cleft repairs.

This randomized controlled trial will be conducted in Cairo hospital (Abu El-Reesh El-Mounira Children University Hospital). To ensure clinical facilities, medical expertise, and target patient access, this study will be conducted in a hospital. The population density of Cairo and prevalence of bilateral alveolar clefts make it ideal for this research . Cairo study sites will be available upon request and documented in the trial.

Interventions All surgical procedures will be conducted under general anesthesia with nasotracheal intubation, and a first-generation cephalosporin will be administered as antibiotic prophylaxis prior to incision. Autogenous bone grafts will be harvested from the anterior iliac crest using a pediatric minimally invasive technique, involving a 2 cm skin incision made 1 cm lateral to the iliac crest, meticulously dissected to preserve soft tissue. pain management strategies will be employed postoperatively to ensure comprehensive pain control and enhance patient comfort throughout the recovery period.

For the alveolar cleft repair, a sulcular incision will be made to develop full thickness mucoperiosteal advancement flaps extending into the cleft, with careful elevation of buccal flaps above the piriform rim. The bone graft will be contoured to fill the defect, ensuring cortical bone contacts the nasal lining and cancellous bone chips fill remaining spaces. Closure will be performed using interrupted sutures, starting with the nasal floor

DETAILED DESCRIPTION:
Research question:

The primary research question that drives this study is: Does the use of prefabricated acrylic splints increase the stability of the premaxilla and enhance soft tissue healing and graft stability in patients with bilateral alveolar clefts? The above research question uses the PICO (Patient, Intervention, Comparison, Outcome) format to ensure clarity, structure, and focus on the most important aspects of the investigation P - Population: Bilateral alveolar cleft patients I - Intervention: Use of prefabricated acrylic splints C - Comparison: in comparison to the control group that did not use acrylic splints O - Outcome: Enhance premaxillary stability vertical and horizontal assessed by (Lateral Cephalometric Analysis (Radiographically), soft tissue healing, and graft stability

Statement of the problem:

Congenital bilateral alveolar clefts affect many patients from diverse backgrounds, impacting their quality of life . These clefts involve separation of the upper jaw from one alveolus to another, often accompanying cleft lip and palate . Both esthetic and functional issues arise due to impacts on speech, feeding, breathing and appearance from childhood onward . Bone grafting is necessary to reconstruct the maxillary anatomy in bilateral alveolar clefts Premaxillary stability is especially crucial, as it influences bone graft incorporation and craniofacial development . Studies report premaxillary mobility still occurs in 20-40% of treated bilateral clefts at one year post-grafting using standard fixation methods . This instability disrupts integration of autogenous bone grafts and impedes future reconstructive care such as orthodontics . While bone grafting aims to reconstruct the maxilla, premaxilla fixation techniques may remain inadequate to guarantee stability. An alternative is needed to optimize patient outcomes for this patient population.

Rationale for conducting the research:

Bilateral alveolar clefts pose significant management challenges, with current treatments like autogenous bone grafting showing instability in up to 40% of cases within a year, risking graft failure and aesthetic issues . Prefabricated acrylic splints may offer a minimally invasive alternative, potentially improving bone graft outcomes and premaxillary stability, crucial for speech, feeding, and respiration . This study evaluates the efficacy of acrylic splinting versus traditional open healing, aiming to enhance patient outcomes and reduce healthcare costs associated with this congenital condition. This research underscores the need for evidence-based, minimally invasive treatments that can improve quality of life and guide clinical practices for managing bilateral alveolar clefts.

Review of literature:

The existing body of literature on bilateral alveolar clefts and their management reflects several inadequacies and gaps in the evidence base. Bilateral alveolar clefts present unique challenges that have not been fully addressed in the literature on cleft lip and palate management . Limited evidence suggests more focused research in this area. The prevailing treatment options for bilateral alveolar clefts predominantly involve surgical bone grafting procedures. These grafting techniques have shown varying success rates, with factors such as graft quality, surgical technique, and premaxillary stability influencing outcomes. However, the specific challenges posed by bilateral alveolar clefts have not been addressed comprehensively in the existing literature. While grafting procedures have undoubtedly improved the lives of countless patients, there remains a need for more targeted interventions that can enhance premaxillary stability and graft success, particularly in the context of bilateral alveolar clefts . The proposed use of prefabricated acrylic splints represents a novel and innovative approach to address these inadequacies. These splints are designed to provide consistent and reliable support to the premaxilla during the critical early phases of healing following grafting procedures. By minimizing premaxillary mobility, they have the potential to enhance graft success rates, improve premaxillary stability, and enhance the overall outcomes of bilateral alveolar cleft repairs.

Explanation for choice of comparators:

, standard bone grafting without acrylic splints is considered the 'gold standard' for treating alveolar clefts. Using normal repair as the comparator allows for a clear assessment of the possible advantages and challenges of incorporating acrylic splints into existing best practices.

7. Objectives:

Aim of the Study The primary aim of this study is to assess the impact of prefabricated acrylic splints on premaxillary stability, soft tissue healing, and graft stability in patients with bilateral alveolar clefts.

Hypothesis:

Null Hypothesis (H0): Bilateral alveolar cleft patients who receive prefabricated acrylic splints have similar premaxillary stability, soft tissue healing, and graft stability.

Alternative Hypothesis (H1): Prefabricated acrylic splints improve premaxillary stability, soft tissue healing, and graft stability in bilateral alveolar cleft patients.

The above hypotheses are neutral and not biased. The study tests these hypotheses to obtain objective and evidence-based conclusions about prefabricated acrylic splints for bilateral alveolar cleft repairs.

8. Trial design: The proposed trial is RCT, the gold standard for assessing intervention efficacy. It will be a parallel group RCT, a commonly controlled comparison of two interventions. Two arms will represent the control and test groups in the trial. This trial aims to determine whether prefabricated acrylic splints are better than no splints in a 1:1 allocation ratio.

Allocation Ratio and Framework:

This RCT has a 1:1 allocation ratio, so the control and test groups will each receive the same number of participants. This balanced allocation ensures equal group sizes, reducing bias and enabling a more robust comparison between the two interventions.

Superiority Trial This RCT is a superiority trial to show that prefabricated acrylic splints improve premaxillary stability, soft tissue healing, and graft stability in bilateral alveolar cleft patients. Superiority trials prove the new intervention works better than the control. In this trial, the null hypothesis (H0) states that the two interventions are similar, while the alternative hypothesis (H1) states that prefabricated acrylic splints are better. A superiority trial is needed to determine if the new intervention improves patient outcomes meaningfully and clinically. It is important to determine if prefabricated acrylic splints improve premaxillary stability, soft tissue healing, and graft success in bilateral alveolar cleft patients. A successful superiority trial could support this intervention in clinical practice, improving patient care and outcomes. A 1:1 allocation ratio reduces allocation bias by balancing the study with equal numbers of participants in each group. This design makes control and test group comparisons clear and robust. This trial will inform clinical practice and build knowledge of bilateral alveolar cleft management.

III. Methods

A) Participants, interventions & outcomes 9. Study settings: This randomized controlled trial will be conducted in Cairo hospital (Abu El-Reesh El-Mounira Children University Hospital). To ensure clinical facilities, medical expertise, and target patient access, this study will be conducted in a hospital. The population density of Cairo and prevalence of bilateral alveolar clefts make it ideal for this research . Cairo study sites will be available upon request and documented in the trial.

10. Eligibility criteria:

A suitable and representative sample will be selected by setting trial participant eligibility criteria. the inclusion and exclusion criteria will consider demographics, disease severity, prior treatment, diagnostics, and other factors. This trial must balance accurately representing the target population with avoiding overly restrictive selection criteria.

Inclusion Criteria

1. Patients diagnosed with bilateral alveolar clefts.
2. Age 8- 12 within the specified range.
3. Willingness to comply with trial requirements.

Exclusion Criteria

1. Patients with allergy use acrylic splints.
2. Severe medical conditions such as mental retardation.
3. Inability to provide informed consent or assent.

   Operator-dependent interventions will have clear eligibility criteria for care providers and centers to ensure consistency in administration. To improve external validity and clinical applicability, the trial will avoid overly restrictive participant selection . To ensure generalizability, trial participants must reflect the diversity of the target population.

11. Interventions

All surgical procedures will be conducted under general anesthesia with nasotracheal intubation, and a first-generation cephalosporin will be administered as antibiotic prophylaxis prior to incision .Autogenous bone grafts will be harvested from the anterior iliac crest using a pediatric minimally invasive technique, involving a 2 cm skin incision made 1 cm lateral to the iliac crest, meticulously dissected to preserve soft tissue. pain management strategies will be employed postoperatively to ensure comprehensive pain control and enhance patient comfort throughout the recovery period.

For the alveolar cleft repair, a sulcular incision will be made to develop full thickness mucoperiosteal advancement flaps extending into the cleft, with careful elevation of buccal flaps above the piriform rim. The bone graft will be contoured to fill the defect, ensuring cortical bone contacts the nasal lining and cancellous bone chips fill remaining spaces. Closure will be performed using interrupted sutures, starting with the nasal floor and followed by oral closure, with a stabilizing horizontal mattress suture for added stability.

Patients will be preoperatively assigned in a 1:1 ratio to receive either a custom-made prefabricated acrylic splint, designed and trimmed using digital software like Mimics for accurate fit and stabilization of the premaxilla , or no splint, allowing for comparison of premaxillary stability between groups. Both groups will follow a standardized postoperative protocol that includes regular follow-up assessments for premaxillary stability, wound healing, and potential complications, using clinical examination and radiographic evaluation. Data collected will be analyzed using statistical methods to compare outcomes between the experimental and control groups, focusing on premaxillary stability as the primary outcome, with wound healing and complications as secondary measures.

12. Outcomes: The trial will evaluate primary, secondary, and other outcomes with specific and measurable units.

The primary outcome should be:

* Premaxillary stability vertical and horizontal assessed by (Lateral Cephalometric Analysis (Radiographically) at 6 months: Perform lateral cephalometric analysis using images generated from Cone Beam Computed Tomography (CBCT) to assess changes in premaxillary position and stability demographically. This radiographic method will help in quantifying any shifts or instability in the premaxilla over time. Soft Tissue Healing: Evaluated based on clinical signs of healing, such as absence of erythema, edema, and wound dehiscence.
* Graft Stability: Radiographic Assessment: Use radiographic techniques, including standard X-rays or CBCT, to evaluate the integration, position, and retention of the bone graft. This will involve checking for signs of graft resorption or failure and measuring overall graft stability over time.

Secondary objectives

* Assessment of Bone Gain and premaxillary stability: Assessed by Cone Beam Computed Tomography (CBCT) Following Periotest Assessment (Clinically): Use the Periotest device to quantitatively measure the mobility and stability of the premaxillary segment. This assessment provides a clinical determination of the segment's stability using specific metrics related to the damping characteristics of the periodontium and bone.

This secondary objective aims to quantitatively analyze the extent of bone regeneration following periodontal treatments using Cone Beam Computed Tomography (CBCT). CBCT is a state-of-the-art imaging technology that provides high-resolution, three-dimensional images of the teeth and jawbones. It is particularly valuable in periodontics for assessing bone structure, detecting defects, and monitoring bone density changes over time.

Prioritization of Outcome Outcome Method of Measurement Unit of Measurement Primary outcome

Premaxillary Stability by (Lateral Cephalometric Analysis (Radiographically) Numerical

Secondary outcome Bone Gain and Premaxilla stability Cone Beam Computed Tomography (CBCT) and Periotest Assessment (Clinically) Numerical

13. Participant timeline A schematic diagram or Gantt chart will be created to provide a clear and concise timeline of the study visits, enrollment process, interventions, and assessments performed on participants. This visual representation will help both participants and investigators understand the study flow.

Table 1: Example template of the recommended content for the schedule of the activities performed on participants.

Figure.Exmple template of recommended content for the schedule of Enrolment interventions, and assessment Study period Enrolment Allocation Post-allocation Close-out Timepoint t1 (Week 1), t2 (Week 2) t0 (Week 3) t3 (Month 1), t4 (Month 3), t5 (Month 6), t6 (Month 9) t Final (Month 12) Enrolment

Eligibility screen t1 (Week 1) Informed consent t2 (Week 2)

Allocation T0 (week 3) Interventions Intervention A: refabricated acrylic splint at t3 (Month 1) Intervention B: No splint at t3 (Month 1)

Assessments

Baseline Variables: Demographics, cleft severity, prior treatments Captured at t0 (Week 3)

Outcome Variables:

Primary: Premaxillary Stability, Soft Tissue Healing, Graft Stability Measured at t5 (Month 6) and t6 (Month 9) Secondary: Bone Gain (assessed by CBCT) at t6, (Month 9) and Periotest Assessment (Clinically)

Other Data Variables: Follow-up assessments for complications, additional clinical and radiographic evaluations additional assessments (t4, Month 3; t5, Month 6)

14. Sample size: The sample size of the present proposed trial will be estimated using clinical and statistical assumptions. The sample size will be calculated using Premaxillary Stability as the primary outcome. Calculations will consider pain score mean, standard deviation, statistical test, significance level (α), and power (1-β). The nature of the study will determine a 20-30% increase for missing data. A reference for assumed outcome values will support sample size calculations. These calculations will be detailed in the trial protocol for transparency and reproducibility.

15. Recruitment:

The trial will employ various strategies to achieve adequate participant enrollment to reach the target sample size. These strategies will include:

• Location: Participants will be recruited from hospitals in Cairo, Egypt, with a high prevalence of patients with bilateral alveolar clefts.

* By Whom: Recruitment will be carried out by trained research personnel, ensuring standardized recruitment procedures.
* When: Recruitment will occur over a specified duration, which will be detailed in the trial protocol.
* How: Recruitment methods will include referrals from healthcare providers, advertising within hospitals, and community outreach programs.
* Expected Recruitment Rates: Anticipated recruitment rates will be established based on the targeted population and historical enrolment data.

B) Assignment of interventions 16. Allocation: 16a. Randomization:

• To randomise participants, the investigator (PI) will utilise the Research Randomizer (https://www.randomizer.org/), which enables completely automatic randomization for various sorts of research.

• A 1:1 ratio of participants will be randomised to both the control and treatment groups.

16b. Allocation concealment mechanism: Allocation will be hidden behind sequentially numbered, opaque, sealed envelopes." An impartial researcher who is not engaged in participant recruitment, data collection, or evaluation will create the envelopes holding the randomized group allocations. At the time of treatment allocation, envelopes will be randomly mixed in a box and picked by participants.

16c. Implementation The principal researcher, who will be working under the supervision of the supervisor, is the one who will be responsible for enrolling participants and assigning people to receive intervention.

17. Masking/blinding:

This is a double-blind experiment for the following reasons:

* To avoid bias in subjective results, participants will be blinded to their treatment allocation.
* To prevent measurement and assessment bias, outcome assessors will likewise be blinded.
* Because the procedures vary across groups, the investigator cannot be blinded.
* Blinding of participants and assessors seeks to increase the objectivity and validity of findings by reducing possible biases.

C) Data collection, management, and analysis:

18. Data collection methods The primary outcome of premaxillary stability will be assessed by blinded, professional orthodontists utilizing standardized cephalometric analysis of radiographs.

Secondary outcomes were analyzed using set up tools and measures by blinded surgeons.

• All data points will be recorded on case report forms.

• For missing data, retention techniques and intention-to-treat analyses will be used.

• Standardised methods, calibrated assessors, validated equipment, and retention techniques will all help to provide a high-quality, comprehensive dataset.

19. Data management: (PI) under the supervision of the main supervisor will do all of these procedures:

* All information will be input online.
* Patient files must be maintained in numerical order and a safe and easily accessible location.
* After the research is completed, all data will be stored for one year.
* The patient's electronic data and scans will be stored on a One drive file to ensure backup and ease of access.

  20. Statistical methods: Statistical analysis will be done later after approval of the board of Oral & Maxillofacial Surgery Department, Faculty of Dentistry - Cairo University.

D) Data monitoring:

21. Monitoring Data monitoring will be the responsibility of the main supervisor. will assess the outcome measurements as well as any potential side effects that may have an impact on the result.

22. Harms

Potential problems:

* Surgical problems associated with bone grafting, such as infection, haemorrhage, and graft failure.
* Problems with splint material include irritation, inflammation, and wound dehiscence.
* Consequences of general anaesthesia

To reduce risks:

* To avoid infection, strict sterile methods and perioperative antibiotics are used.
* Close monitoring for bleeding problems and meticulous haemostasis
* Splint design and material selection must be meticulous to avoid irritation.
* Anaesthesia is delivered by a professional staff in accordance with procedure.

To keep monitoring of potential risks:

* At follow-ups, participants were checked for symptoms of infection, haemorrhage, and graft problems.
* At each appointment, splint tolerance and wound healing are evaluated.
* Adverse incidents are reported on case report forms and tracked until they are resolved.
* Any major adverse occurrences will be reviewed by a data safety monitoring board.

  23. Audit second supervisor will be the one to do the auditing of the research design.

IV. Ethics and dissemination 24. Research ethics approval The Ethics Committee of Scientific Research of the Faculty of Dentistry at Cairo University is going to review both this protocol and the informed consent form template.

25. Protocol amendments Any changes to the protocol that have an impact on the study's conduct, potential benefit to the patient, or patient safety, such as changes in study objectives, study design, sample sizes, study procedures, or significant administrative aspects, will necessitate a formal amendment to the protocol. The Council of the Department of Oral and Maxillofacial Surgery will approve on such a change.

26. Informed consent The principal investigator (PI) will describe the study's specifics and risks/benefits to interested participants. There will also be full explanation Prior to enrolling, participants will have the option to interact with researchers and ask questions.

Before enrolling, willing individuals will provide written informed permission. There will be consent forms accessible in Arabic. (mother language of the participants).

27. Confidentiality How personal information about enrolled participants will be collected, shared, and maintained in order to protect confidentiality before, during, and after the trial.

28. Declaration of interest The study is self-funded and there is no conflict of interest to declare.

29. Access to data The data sets will be available to the whole study team. Password protection will be applied to all data sets. To protect confidentiality, all identifying participant information will be removed from data sent to project team members, and the participant will only be identified by patient number.

30. post-trial care In the case of an emergency, all patients will be given the principal research contact number.

The monitoring will continue until all of the patients are happy.

31. Dissemination policy

* The findings of the study will be published as part of the prerequisites for a master's degree in oral and maxillofacial surgery.
* Topics for presentation or publishing will be offered to the author as well.
* The finding of the study will be presented in international conferences.
* Display findings at community centres, public libraries, and town halls.

EndNote Version 20

Our proposed study relies on EndNote version 20 for reference management and citation and bibliography accuracy. This software streamlines research by organizing the extensive library of academic materials on alveolar cleft bone graft repairs. A key function of EndNote is managing and categorizing references. Researchers can organize research articles, studies, and other academic resources. This feature is essential for organizing relevant literature for a complex study. Additionally, EndNote simplifies citation and bibliography creation. Research team collaboration is encouraged by the software. EndNote simplifies reference sharing for interdisciplinary studies like this, making it easier for researchers to collaborate.

V. Appendices 32. Informed consent

consent forms and other related documentation will be given to the participant's guardian. These will be fully explained, including details about the procedure, the intervention, and possible complications.

ELIGIBILITY:
Eligibility criteria:

A suitable and representative sample will be selected by setting trial participant eligibility criteria. Mesa et al (2016) claimed that, the inclusion and exclusion criteria will consider demographics, disease severity, prior treatment, diagnostics, and other factors. This trial must balance accurately representing the target population with avoiding overly restrictive selection criteria.

Inclusion Criteria

1. Patients diagnosed with bilateral alveolar clefts.
2. Age 8- 12 within the specified range.
3. Willingness to comply with trial requirements.

Exclusion Criteria

1. Patients with allergy use acrylic splints.
2. Severe medical conditions such as mental retardation.
3. Inability to provide informed consent or assent.

Operator-dependent interventions will have clear eligibility criteria for care providers and centers to ensure consistency in administration. To improve external validity and clinical applicability, the trial will avoid overly restrictive participant selection (Sessler & Imrey 2015; Aggarwal & Ranganathan 2019). To ensure generalizability, trial participants must reflect the diversity of the target population.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome should be: Premaxillary stability vertical and horizontal assessed by (Lateral Cephalometric Analysis (Radiographically) at 6 months: Perform lateral cephalometric analysis using images generated from Cone Beam Computed Tomography ( | 6 MONTHS
  Primary Outcome Measure:
  Outcome Measure Name: Premaxillary Stability Description: Assess the stability of the premaxilla both vertically and horizontally.
  Assessment Method: Lateral Cephalometric Analysis using images from Cone Beam Computed Tomography (CBCT).
  Time Frame: 6 months post-procedure. Units of Measure: Stability will be quantified in millimeters (mm) for both vertical and horizontal displacements.

SECONDARY OUTCOMES:
Secondary Outcome Measures: Outcome Measure Name: 1) Soft Tissue Healing 2) Outcome Measure Name: Graft Stability | 6 MONTHS
  Secondary Outcome Measures:
  Outcome Measure Name: Soft Tissue Healing Description: Evaluate the healing of soft tissues surrounding the surgical site.
  Assessment Method: Clinical examination to assess signs such as erythema, edema, and wound dehiscence.
  Time Frame: At 1 week, 1 month, 3 months, and 6 months post-procedure. Units of Measure: Healing status categorized qualitatively as healed, healing, or not healed.
  Outcome Measure Name: Graft Stability Description: Determine the integration and stability of the bone graft. Assessment Method: Radiographic evaluation using X-rays or CBCT. Time Frame: 6 months post-procedure. Units of Measure: Stability reported qualitatively based on radiographic evidence

OTHER OUTCOMES:
Stability will be quantified in millimeters (mm) for both vertical and horizontal displacements. | 6 MONTHS
  Stability will be quantified in millimeters (mm) for both vertical and horizontal displacements.

IPD SHARING:
Plan to Share IPD: Undecided